CLINICAL TRIAL: NCT03379909
Title: Phase II Study of Oral Metformin for Intravesical Treatment of Non-muscle-invasive Bladder Cancer
Acronym: TROJAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, J.W. Wilmink, Medical Oncologist, Associate Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Medonc-17-11
Record Dates: First submitted 2017-12-16; First posted 2017-12-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Superficial Bladder Cancer; Bladder Cancer
Keywords: metformin; marker lesion
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Metformin orally at doses up to 1500 mg twice daily for 3 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin orally at doses up to 1500 mg twice daily for 3 months.

SUMMARY:
A multi-center, open-label, phase II clinical study of metformin in up to evaluable 49 patients with low-grade NMIBC with the aim to determine the overall response to administration of oral metformin for 3 months in a index papillary NMIBC tumour.

DETAILED DESCRIPTION:
A multi-center, open-label, phase II clinical study of metformin in up to 49 patients with low-grade NMIBC with the aim to determine the overall response to administration of oral metformin for 3 months in a index tumour (0.5-1 cm) selected ane measured during cystoscopy. All patients will receive metformin orally at doses up to 1500 mg twice daily. Metformin treatment will start directly after informed consent is obtained. After 3 months of metformin treatment, the effect of metformin on the index lesion is evaluated by performing a transurethral resection of the bladder tumour under anaesthesia. Residual tumour, if present at this evaluation, will be resected. In case of complete disappearance of the index lesion the former tumour area will be biopsied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients with primary or recurrent suspectedTa or T1, G1 or G2 (low grade) urothelial carcinoma of the bladder with no suspicion of carcinoma in situ.
* Patients must have at least 1 lesion but no more than 5.
* There must be one index lesion measuring between 0.5 and 1.0 cm in its greatest dimension.
* Bimanual examination immediately following cystoscopyshould be carried out and no mass should be felt.
* Adequate renal function (eGFR >50 ml/min/1.73m2 according to CKD-EPI). (47)
* Adequate liver function (bilirubin <1.5 times upper limit of normal, ALAT or ASAT <2.5 the upper limit of normal).
* Eligible patients must be fully informed of the investigational nature of the study and written signed informed consent must be obtained prior to any study specific investigations.
* Mentally, physically, and geographically able to undergo treatment and follow up.

Exclusion Criteria:

* Patients with positive cytology (suspected for high-grade urothelial carcinoma, TPS 4 or TPS 5) or suspected grade 3 tumours.
* Patients with diabetes mellitus receiving metformin or having received metformin in the past 6 months.
* Patients who have received intravesical treatment (chemotherapy or immunotherapy) within the last 3 months.
* Patients that are currently receiving other anti-cancer therapy.
* Patients with existing urinary tract infection or recurrent severe bacterial cystitis.
* Patients that need to be treated with a transurethral catheter.
* Patients with urogenital tumours with histology other than urothelial carcinoma (i.e. squamous cell or adenocarcinoma) or with urothelial carcinoma involving the upper tract or the prostatic urethra.
* Patients with a history of other primary malignancy (other than squamous or basal cell skin cancers or cone biopsied CIS of the uterine cervix or prostate carcinoma treated curatively with normal PSA values at inclusion) in the last five years.
* Patients with active, uncontrolled impairment of the renal, hepatobiliary, cardiovascular, gastrointestinal, urogenital, neurologic or hematopoietic systems that, in the opinion of the investigator, would predispose to the development of complications from the administration of metformin.
* Patients who are using loop diuretics, cimetidine, ranitidine, cetirizine, trimethoprim, vandetanib, kinidine and/or HIV medication, for which no reasonable alternative is available.
* Women who are pregnant or lactating. Individuals of reproductive potential may not participate unless agreeing to use an effective contraceptive method for themselves and/or their sexual partner.
* Patients with ECOG-WHO performance status of 3 or 4.
* Patients with a known history of alcohol abuse.
* Patients with a known hypersensitivity to metformin.
* Patients who in the investigator's opinion, cannot comply with provisions of the protocol or do not understand the nature of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall response | 3 months
  The primary outcome is the objective response rate (complete responses) after 3 months of treatment with metformin. Evaluable patients are those who have received at least 500 mg metformin twice daily for one week and who undergo a cystoscopy for marker lesion removal.

SECONDARY OUTCOMES:
Time to recurrence | 5 years
  The duration of the time to recurrence of NMIBC after stopping metformin treatment. Patients will be followed for a maximum duration of 5 years.
Toxicity of metformin treatment | 3 months
  The number of grade 1-4 and grade 5 (fatal) NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE) events during treatment with metformin. All patients will be evaluable for toxicity from the time of their first treatment with metformin.
Partial response | 3 months.
  At least 30% reduction in the longest diameter of the marker lesion.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - RadboudUMC, Nijmegen, Gelderland
  - Sint Franciscus Gasthuis, Rotterdam, South Holland
  - Academic Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molenaar RJ, van Hattum JW, Brummelhuis IS, Oddens JR, Savci-Heijink CD, Boeve ER, van der Meer SA, Witjes JF, Pollak MN, de Reijke TM, Wilmink JW. Study protocol of a phase II clinical trial of oral metformin for the intravesical treatment of non-muscle invasive bladder cancer. BMC Cancer. 2019 Nov 21;19(1):1133. doi: 10.1186/s12885-019-6346-1. PMID 31752752